CLINICAL TRIAL: NCT01774851
Title: Randomized, Open Label, Phase 2 Study of MM-111 and Paclitaxel With Trastuzumab in Patients With HER2 Positive Carcinomas of the Distal Esophagus, Gastroesophageal (GE) Junction and Stomach Who Have Failed Front Line Metastatic or Locally Advanced Therapy
Brief Title: A Study of MM-111 and Paclitaxel With Trastuzumab in Patients HER2 Positive Carcinomas of the Distal Esophagus, Gastroesophageal (GE) Junction and Stomach
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMB recommendation due to lack of efficacy. There were no safety signals.
Sponsor: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-111-13-02-04
Record Dates: First submitted 2013-01-10; First posted 2013-01-24 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: HER-2 Gene Amplification; Esophagus Cancer; Gastroesophageal Junction Cancer; Stomach Cancer
Keywords: HER-2 Gene Amplification; Esophagus Cancer; Gastroesophageal Junction Cancer; Stomach Cancer; Her2 Positive; Her2+; Esophageal Cancer; Metastatic
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasm Metastasis | interventions — MM-111; Paclitaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1a (Experimental): MM-111 + Paclitaxel + Trastuzumab
  Interventions: Drug: MM-111; Drug: Paclitaxel; Drug: Trastuzumab
- Arm 1b (Active Comparator): Paclitaxel + Trastuzumab
  Interventions: Drug: Paclitaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: MM-111 — MM-111 (IV)
  Arms: Arm 1a
Drug: Paclitaxel — Paclitaxel (IV)
Drug: Trastuzumab — Trastuzumab (IV)

SUMMARY:
To determine whether the combination of MM-111 plus paclitaxel and trastuzumab is more effective than paclitaxel and trastuzumab alone

DETAILED DESCRIPTION:
This is a randomized, open Label, Phase 2 Study of MM-111 and Paclitaxel withTrastuzumab in Patients with HER2 Positive Carcinomas of the Distal Esophagus, Gastroesophageal (GE) Junction and Stomach Who Have Failed Front Line Metastatic or Locally Advanced Therapy. Approximately 120 patients will be randomized in a 1:1 ratio between the experimental and comparator arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have documentation of histologically or cytologically confirmed metastatic or locally advanced adenocarcinoma of the distal esophagus, GE junction or stomach
* Patients must have documentation of histologically or cytologically confirmed HER2 expression
* Patients must be ≥18 years of age
* Patients must have ECOG PS of 0, 1, or 2
* Patients must have adequate hematologic status, renal and hepatic function

Exclusion Criteria:

* Patients with known hypersensitivity to any of the components of MM-111
* Patients with a known history of hypersensitivity to paclitaxel or other drugs formulated in Cremophor® EL
* Patients with a known history of hypersensitivity to trastuzumab or any of its components (group 1 patients only)
* Patients with an active infection or with an unexplained fever >38.5°C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-01; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akos Czibere, MD, PhD, Study Director — Merrimack Pharmaceuticals
Locations (19):
- United States (19):
  - Birmingham, Alabama
  - Los Angeles, California
  - Stanford, California
  - Denver, Colorado
  - Ocala, Florida
  - St. Petersburg, Florida
  - Urbana, Illinois
  - Boston, Massachusetts
  - Rochester, Minnesota
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Buffalo, New York
  - Durham, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Paclitaxel + Trastuzumab
- Experimental Group: MM-111 + trastuzumab + paclitaxel
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Trastuzumab + paclitaxel
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Median (Full Range); unit: years] | 62.5 [35 to 81] | 63.5 [31 to 78] | 63 [31 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 40 | 37 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 41 | 41 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 30 | 29 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26
  Denmark | 0 | 1 | 1
  France | 1 | 0 | 1
  Korea, Republic of | 11 | 10 | 21
  Spain | 9 | 8 | 17
  Taiwan | 2 | 2 | 4
  United Kingdom | 6 | 8 | 14
Subject of child bearing potential [Count of Participants; unit: Participants] | 0 | 2 | 2
Height [Median (Full Range); unit: cm] | 172 [154.2 to 190.5] | 170.19 [152.4 to 193.0] | 171 [152.4 to 193]
Weight [Median (Full Range); unit: kg] | 73.97 [47.1 to 126.6] | 68 [41.2 to 98.2] | 72.51 [41.2 to 126.6]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Target and non-target lesion antitumor response and disease progression during treatment with each dosing regimen will be evaluated using the international criteria proposed by the RECIST v1.1. Disease status will be assessed every 8 weeks from the date of the first dose of any drug in a regimen.
Time Frame: 30 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 42 | 42
weeks | 23.3 [12.1 to 27.0] | 9.6 [8.0 to 15.7]

ADVERSE EVENTS:
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 18/42 | 11/42
Serious Adverse Events (participants affected / at risk) | 16/42 | 19/42
Other Adverse Events (participants affected / at risk) | 26/42 | 39/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=42) | Experimental Group (N=42)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper GI haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
GI obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Blood cortisol decreased (Investigations) | 1 (1) | 0 (0)
Transaminase increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Pleural effusion (General disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=42) | Experimental Group (N=42)
Diarrhoea (Gastrointestinal disorders) | 12 (12) | 22 (22)
Nausea (Gastrointestinal disorders) | 11 (11) | 11 (11)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6)
Vomiting (Gastrointestinal disorders) | 5 (5) | 13 (13)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 9 (9) | 14 (14)
Asthenia (General disorders) | 8 (8) | 7 (7)
Oedema peripheral (General disorders) | 7 (7) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 17 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2) | 5 (5)
Peripheral sensory neuropathy (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 4 (4)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Neurotoxicity (Nervous system disorders) | 3 (3) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 14 (14) | 15 (15)
Neutropenia (Blood and lymphatic system disorders) | 7 (7) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 18 (18)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Neutrophil count decreased (Investigations) | 4 (4) | 8 (8)
Weight decreased (Investigations) | 2 (2) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Conjunctivitis (Eye disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Following the recommendation of the data monitoring committee, this study was terminated prior to enrollment being completed due to lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No